CLINICAL TRIAL: NCT04359667
Title: Prognostic Value of Serum Interleukin-6 (IL-6) and Soluble Interleukin-6 Receptor (sIL-6R) in Severe Coronavirus Disease (COVID-19) Pneumonia Treated With Tocilizumab - a Prospective Single Center Study (UHID-COVID19)
Brief Title: Serum IL-6 and Soluble IL-6 Receptor in Severe COVID-19 Pneumonia Treated With Tocilizumab
Acronym: UHID-COVID19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital for Infectious Diseases, Croatia (Other)
Responsible Party: Sponsor
Other Study IDs: UHID-04
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; Severe Pneumonia
Keywords: COVID-19; severe pneumonia; Interleukin-6; tocilizumab
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- tocilizumab: one infusion of TCZ 8 mg/kg i.v., with a maximum dose of 800 mg, and SOC treatment according to local guidelines (hydroxychloroquine or/and lopinavir/ritonavir or/and remdesivir).
  Interventions: Drug: Tocilizumab 20 MG/ML Intravenous Solution [ACTEMRA]

INTERVENTIONS:
Drug: Tocilizumab 20 MG/ML Intravenous Solution [ACTEMRA] — 1 - 8 mg per kg of body weight once, maximal 800 mg per dose (can be repeated once more after 12 hours, per clinician's assessment)
  Other Names: RoActemra, Anatomical Therapeutic Chemical (ATC) Code L04AC07

SUMMARY:
This is a single arm, prospective, observational, single center study to assess the role of interleukin-6 (IL-6) and soluble interleukin 6 receptor (sIL-6R) as predictors of efficacy and safety outcomes in patients with severe coronavirus disease (COVID-19) pneumonia treated with tocilizumab. At least 30 patients will be enrolled who are diagnosed with severe COVID-19 pneumonia and meet the entry criteria.

DETAILED DESCRIPTION:
Patients must be at least 18 years of age with severe COVID-19 pneumonia (and/or ARDS) confirmed per World Health Organization (WHO) criteria, and evidence of pulmonary infiltration (by chest X-ray and/or CT scan), including a virological confirmation of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection by positive polymerase chain reaction (PCR) of any specimen; e.g., respiratory, blood, urine, stool, other bodily fluid.

At the time of enrollment, patients have to fulfill criteria of the local recommendations for the treatment with tocilizumab (TCZ): hypoxemia (defined as arterial oxygen partial pressure/fraction of inspired oxygen (PaO2/FiO2) ratio ≤300 mmHg and/or peripheral capillary oxygen saturation (SpO2) ≤93%) regardless of the oxygenation method including low-flow oxygen administration on nasal cannula or mask with oxygen flow rate of > 12 liters per minute, high-flow oxygen through nasal cannula, noninvasive ventilation (NIV) whatever the modalities of ventilation, invasive ventilation through tracheal intubation or tracheostomy, and extracorporeal oxygenation, despite being on standard of care (SOC), which may include anti-viral treatment, low dose steroids, antimalarials and supportive treatment and care.

Patients in whom, in the opinion of the treating physician, progression to death is imminent and inevitable within the next 24 hours, will be excluded from the study. Patients with active tuberculosis (TB) or suspected active bacterial, fungal, viral, or other infection (besides COVID-19) will be excluded from the study.

Patients will receive one infusion of TCZ 8 mg/kg i.v., with a maximum dose of 800 mg, and SOC treatment according to local guidelines (hydroxychloroquine or/and lopinavir/ritonavir or/and remdesivir).

If the clinical signs or symptoms worsen or do not improve (reflected by sustained fever or at least a one-category worsening on the 7-category ordinal scale of clinical status), one additional infusion of blinded treatment of TCZ or placebo may be given, after more than 12 hours per local protocol.

The study assessments to be conducted include the following: physical examination, vital signs, oxygen saturation, assessment of consciousness, presence and absence of respiratory support, adverse events, concomitant therapies, clinical laboratory tests, and nasopharyngeal swabs.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form by any patient capable of giving consent, or, when the patient is not capable of giving consent, by his or her legal/authorized representative
* Age ≥18years at time of signing Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgment
* Hospitalized due to severe COVID-19 pneumonia (and/or ARDS) confirmed per World Health Organization criteria, and evidence of pulmonary infiltration (by chest X-ray and/or CT scan), including a virological confirmation of SARS-CoV-2 infection by positive PCR of any specimen; e.g., respiratory, blood, urine, stool, other bodily fluid
* Hypoxemia (defined as a PaO2/FiO2 ratio ≤300 mmHg and/or SpO2≤93%) regardless of their oxygenation device (including low-flow oxygen administration on nasal cannula or mask with oxygen flow rate of > 12 liters per minute), high-flow oxygen through nasal cannula, noninvasive ventilation (NIV) whatever the modalities of ventilation, invasive ventilation through tracheal intubation or tracheostomy, and extracorporeal oxygenation, despite being on SOC, which may include anti-viral treatment, low dose steroids, and supportive care

Exclusion Criteria:

* Known severe allergic reactions to TCZ or other monoclonal antibodies
* Active TB infection
* Suspected active bacterial, fungal, viral, or other infection (besides COVID-19)
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments
* Have received oral anti-rejection or immunomodulatory drugs (including TCZ) within the past 6 months
* alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >10 times the upper limit of the normality detected within 24 hours at screening or at baseline
* absolute neutrophil count (ANC) <1000/µL at screening and baseline
* Platelet count <50,000/µL at screening and baseline
* Pregnant or breastfeeding, or positive pregnancy test in a pre-dose examination
* Any serious medical condition or abnormality of clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 yrs with severe COVID-19 pneumonia (and/or ARDS) confirmed per WHO criteria, and evidence of pulmonary infiltration (by chest X-ray and/or CT scan), including a virological confirmation of SARS-CoV-2 infection by PCR of any specimen; e.g., respiratory, blood, urine, stool, other bodily fluid. At enrollment, patients have to fulfill criteria of local recommendations for tocilizumab treatment: hypoxemia regardless of the oxygenation method including low-flow oxygen administration on nasal cannula or mask with oxygen flow rate of > 12 liters per minute, high-flow oxygen through nasal cannula, noninvasive ventilation whatever the modalities of ventilation, invasive ventilation through tracheal intubation or tracheostomy, and extracorporeal oxygenation, despite being on SOC, which may include anti-viral treatment, low dose steroids, antimalarials and supportive treatment and care.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-04-16 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
serum interleukin-6 and soluble interleukin-6 receptor as biomarkers of clinical outcomes in patients with severe coronavirus disease (COVID-19) pneumonia treated with tocilizumab | baseline
  to evaluate the role of laboratory markers as predictors of survival in severe COVID-19 pneumonia patients treated with tocilizumab
serum interleukin-6 and soluble interleukin-6 receptor as biomarkers of clinical outcomes in patients with severe coronavirus disease (COVID-19) pneumonia treated with tocilizumab | 24 hours post treatment
  to evaluate the role of laboratory markers as predictors of survival in severe COVID-19 pneumonia patients treated with tocilizumab
serum interleukin-6 and soluble interleukin-6 receptor as biomarkers of clinical outcomes in patients with severe coronavirus disease (COVID-19) pneumonia treated with tocilizumab | 48 hours post treatment
  to evaluate the role of laboratory markers as predictors of survival in severe COVID-19 pneumonia patients treated with tocilizumab
serum interleukin-6 and soluble interleukin-6 receptor as biomarkers of clinical outcomes in patients with severe coronavirus disease (COVID-19) pneumonia treated with tocilizumab | on Day 7
  to evaluate the role of laboratory markers as predictors of survival in severe COVID-19 pneumonia patients treated with tocilizumab
serum interleukin-6 and soluble interleukin-6 receptor as biomarkers of clinical outcomes in patients with severe coronavirus disease (COVID-19) pneumonia treated with tocilizumab | on Day 28
  to evaluate the role of laboratory markers as predictors of survival in severe COVID-19 pneumonia patients treated with tocilizumab

CONTACTS AND LOCATIONS:
Overall Officials: Rok Civljak, MD, PhD, Principal Investigator — University Hospital for Infectious Diseases "Dr Fran Mihaljevic"
Locations (1):
- University Hospital for Infectious Diseases "Dr Fran Mihaljevic", Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided